CLINICAL TRIAL: NCT04024527
Title: Efficacy of High Dose of Dual Therapy Plus Metronidazole for Helicobacter Pylori Rescue Treatment: A Randomized Clinical Trial
Brief Title: High Dose of Dual Therapy Plus Metronidazole for Helicobacter Pylori RescueTreatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjyy20190715
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual therapy (Active Comparator): Esomeprazole 40mg bid and Amoxicillin 1.0g tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin
- Metronidazole plus dual therapy (Experimental): Esomeprazole 40mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Metronidazole

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Metronidazole — Antibiotic for H. pylori eradication
  Arms: Metronidazole plus dual therapy

SUMMARY:
Dual therapy containing high dose of proton pump inhibitor (PPI) and amoxicillin had showed excellent eradication results with Helicobacter pylori first-line treatment. However, no study has examined the the efficacy of high dose of dual therapy or dual therapy plus metronidazole for H. pylori rescue treatment.This study is designed to evaluate the efficacy and safety of the addition of metronidazole to high dose of dual therapy for H. pylori rescue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with previous treatment failure

Exclusion Criteria:

* Less than 18 years old or older than 80 years
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth,antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value)

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D.,Ph.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding ZH, Huang Y, Chen JN, Luo LS, Zhang W, Liang X, Lu H. A randomized superiority clinical trial: metronidazole improved the efficacy of high-dose dual therapy in Helicobacter pylori rescue treatment. J Antimicrob Chemother. 2023 Mar 2;78(3):828-831. doi: 10.1093/jac/dkad020. PMID 36719104